CLINICAL TRIAL: NCT03025061
Title: Within-day and Between-day Repeatability of the Breath Pattern in Healthy Children and in Children With Moderate Asthma
Brief Title: Within-day and Between-day Repeatability of the Breath Pattern in Healthy Children and in Children With Asthma
Acronym: CERS
Status: Completed | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 5/2016
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Asthma; Healthy
Keywords: Breath pattern; Children; Repeatability
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 15 children with moderate asthma: Assessment of E-nose measurements: three E-nose measurements on 15 children with moderate asthma (of both sex and 6-11 years old): first measurement, second one after 30 minutes, third one after 7 days. These children attend the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (IBIM CNR).
  Interventions: Other: Assessment of E-nose measurements
- 30 healthy children: Assessment of E-nose measurements: three E-nose measurements on 30 healthy children (of both sex and 6-11 years old): first measurement, second one after 30 minutes, third one after 7 days. These children attend the primary schools involved in the municipal project "Educational Pathways" (Palermo).
  Interventions: Other: Assessment of E-nose measurements

INTERVENTIONS:
Other: Assessment of E-nose measurements — Breath sampling through E-nose pneumopipe

SUMMARY:
"Within-day and Between-day Repeatability of the Breath Pattern in Healthy Children and in Children With Moderate Asthma" is an observational prospective study in outpatient clinic of Pediatric Allergology & Pulmonology (PAP) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (IBIM CNR), Italy.

The electronic nose (E-nose) has been proposed as a novel, non-invasive tool to evaluate the level of airway inflammation for different respiratory diseases, especially in children. To date, there are no data on the within-day and the between-day repeatability of the breath pattern in healthy children and in children with moderate asthma.

The breath pattern will be analyzed by collecting, for each child, three samples of the breath through the E-nose. Within-day repeatability will be assessed using two consecutive measurements (the second one after 30 minutes). Between-day repeatability will be assessed using a third measurement repeated after 7 days.

The study is expected to provide information about the accuracy of E-nose measurements for a child population.

ELIGIBILITY:
The inclusion criteria for asthmatic children are:

1. Moderate asthma (GINA 2015);
2. Age 6-11 years;
3. No upper airway respiratory infections or exacerbations in the last 4 weeks;
4. Steroid-naive asthma;
5. Positive bronchodilator response;
6. Non smoker.

The inclusion criteria for healthy children are:

1. Age 6-11 years;
2. No upper airway respiratory infections in the last 4 weeks;
3. Non smoker;
4. No history of asthma and respiratory diseases during the life;
5. Negative bronchodilator response.

The exclusion criteria are:

1. Symptoms of acute respiratory infection;
2. Immunological and metabolic systemic disease;
3. Major malformations of the upper airways;
4. Active smoker.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A study population of 15 asthmatic children (moderate asthma) attending the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (IBIM CNR).
  A control group of healthy children (n=30), recruited from the primary schools involved in the municipal project "educational pathways" (Palermo, Italy) to which the PAP group partecipates.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Electronic nose measurements | 1 week
  Several volatile organic compounds, including isoprene, 1,2-pentadiene, acetone, ethanol, pentane and ethane, identified in exhaled breath.

SECONDARY OUTCOMES:
Fraction of Exhaled Nitric Oxide (FeNO) | 1 week
Pulmonary function (FEV1, FVC, etc.) | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fasola S, Ferrante G, Sabatini A, Santonico M, Zompanti A, Grasso S, Antonelli Incalzi R, La Grutta S. Repeatability of exhaled breath fingerprint collected by a modern sampling system in asthmatic and healthy children. J Breath Res. 2019 May 1;13(3):036007. doi: 10.1088/1752-7163/ab1765. PMID 30965288